CLINICAL TRIAL: NCT04901949
Title: Comparison of the Severity and Complications of Acute Pancreatitis in Obese and Non-obese Patients According to the Atlanta and Balthazar Scores
Brief Title: The Course of Acute Pancreatitis in Patients With Different BMI Groups
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: Aa654321+
Record Dates: First submitted 2021-05-03; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Acute Pancreatitis; Obesity; Body Weight
Keywords: Acute pancreatitis; Obesity; Body Mass Index; Revised Atlanta Scoring; Balthazar Scoring
MeSH Terms: conditions — Pancreatitis; Obesity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BMI Group 1: If BMI is less than 24,9 kg/m2
- BMI Group 2: If BMI is between 25 - 30 kg/m2
- BMI group 3: If BMI is more than 30,1 kg/m2

SUMMARY:
In obese (OB) patients, the presence of an increased inflammatory state in the body due to the increase in abdominal adipose tissue and increase in the frequency of gallstones and lipid levels are expected to increase the development of acute pancreatitis (AP). The effect of obesity on the clinical course of acute pancreatitis has much been attracted the attention of researchers.

The aim of this study is to evaluate whether the prevalence and severity of AP, as well as Balthazar tomographic scoring, differs in BMI groups (normal, overweight, obese).

DETAILED DESCRIPTION:
Today, the incidence of acute pancreatitis (AP) is gradually increasing. According to the Atlanta criteria, the presence of two of the three findings (characteristic abdominal pain starting from the epigastrium and spreading to the left upper quadrant in a belt manner from there, which is severe enough to bring the patient to the emergency room, amylase and lipase values being 3 of normal, radiological imaging being compatible with AP) is sufficient for the diagnosis. The disease has a mild course of 80% of patients and usually resolves within a week, but the course is severe enough to require intensive care treatment in 15-20% of patients. AP may have local (pseudocyst, abscess, necrosis, vascular thrombosis) and systemic (organ failure; lung, heart, gastrointestinal, and renal) complications.

The frequency of obesity (OB) is also increasing in societies, according to the world health organization (WHO) data, 39% of women aged ≥18 and 39% of men were overweight in 2016 in the world. Overweight and OB are defined as excessive fat accumulation that can impair health, which is an important risk factor for many chronic diseases, including diabetes, cardiovascular disease, and cancer. While once seen only as a problem in high-income countries, overweight and OB are increasing significantly in low- and middle-income countries. Body mass index (BMI) is a simple index commonly used to classify overweight and OB in adults. It is defined by dividing a person's weight by the square of their height (kg/m2). According to WHO, if the BMI is between 25-30 kg/m2, it is considered overweight, if it is ≥30,1 kg/m2, it is considered OB. An increase in the frequency of gallstones, in lipids, and in abdominal adipose tissue in OBs are expected to increase the development of AP as the cytokine and tumor necrosis factor (TNF)-α levels in the body increase. In recent years, the number of publications indicating a relationship between OB and AP frequency has been increasing.

Retrospectively, 1550 patients who followed up at the Gastroenterology Clinic of Bezmialem Vakif University between 10/2010 and 02/2020, aged ≥18 years and diagnosed with AP according to the Atlanta definition criteria were screened. After the exclusion of patients with incomplete data, 1334 patients were included in the study.

Patients' age, gender, smoking/alcohol usage, presence of diabetes/hypertension, and etiologies that cause AP and BMI were recorded.

The patients were divided into 3 groups according to their BMI;

* Group 1 (non-obese; normal) [BMI ≤ 24,9 kg/m2: n: 302: 152 ♂, 150]
* Group 2 (overweight) [BMI 25-30 kg/m2: n: 500: 262♂, 238♀]
* Group 3 (obese) [BMI> 30.1kg/m2: n: 532; 200♂, 332♀]. As of laboratory tests; Leukocyte number (n: 4.5-11x100/microliter), hematocrit (n: 35.5-48%), C reactive protein (CRP) (n: 0-5mg / dl), blood urea nitrogen (BUN) ( n: 9.8-20.1mg / dL), serum creatinine (n: 0.57-1.11mg / dl)] levels.

As of radiologic evaluation, Balthazar tomographic scoring; [scores are grouped as mild (scores 0-3), moderate (scores: 4-6), severe (scores 7-10), and scores are defined as 0:normal, 1:increase in pancreatic size, 2:inflammatory changes in pancreatic tissue, and peripancreatic fatty tissue, 3:irregularly bordered, single fluid collection, 4:irregularly circumscribed 2 or more fluid collections, with various degrees of necrosis levels between 5 and 10].

And revised Atlanta scores; A) mild AP: no organ insufficiency and local complications B) moderate AP; the presence of local complications and transient organ insufficiency (<48h) C) severe AP: permanent organ insufficiency (> 48h)] Complications (0: absent 1: local complications 2: systemic complications 3: mixed serious complications/comorbid conditions 4: infectious-sepsis) Need for the interventional procedures such as endoscopic retrograde cholangiopancreatography (ERCP) and endosonography (EUS) Length of hospital stay (in days) Need for the intensive care unit hospitalization The number of AP attacks in the future after discharge was recorded.

Statistical Analysis

Descriptive statistics of the obtained data were calculated as Mean +/- (standard deviation) (SD), minimum, maximum, percentiles (25th, median, and 75th), and frequencies (count and percent), depending on the type of variables. The consistency and relationships between BMI groups, Balthazar scores, and Atlanta scores were analyzed using Kappa statistics and Kendall Tau-b statistics. The compliance of numerical properties to the normal distribution was examined using the Shapiro-Wilks test. One-Way ANOVA model, one of the univariate analyzes, was used to compare BMI groups and Atlanta score groups in terms of numerical features, significant differences were determined by the posthoc Tukey test. Relationships between categorical features and BMI groups and Atlanta scores were analyzed using the Pearson Chi-Square test. In addition, the combined effects of the measured features on exitus, ICU hospitalization status, and hospitalization time over 11 days were re-examined with multivariate logistic regression analysis, and in this analysis, the properties whose effects were not significant were removed from the model with the Backward variable selection method. Statistical significance level was accepted as P <= 0.05 and Statistical Package for the Social Sciences program (SPSS) (ver. 23) program was used in calculations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pancreatitis diagnosis according to the revised Atlanta criteria.

Exclusion Criteria:

* Patients who sign a treatment rejection form immediately after admission to the hospital and leave the hospital,
* Psychiatric patients
* Patients with very poor general conditions will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of acute pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 1334 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The course of acute pancreatitis (mild, moderate, and severe) will be evaluated in patients with different body mass index groups. | Within a month
  The course of acute pancreatitis is defined as mild (no organ insufficiency and local complications), moderate (presence of local complications +/- transient organ insufficiency less than <48h), and severe (permanent organ insufficiency longer than 48h) according to the revised Atlanta scoring. Body mass index is calculated by dividing the weight of a patient (as a kilogram) by the height (as a square meter). Normal weighted patients form Group 1 (≤24,9 kg/m2), overweighted patients form Group 2 (25-30 kg/m2), and obese patients form Group 3 (≥30,1 kg/m2).
Efficacy of acute pancreatitis tomographic scoring (Balthazar) in different body mass index groups | Within a month
  Does the course of acute pancreatitis in the body mass index groups (Group 1, 2, and 3) show parallelism with the tomographic scoring? Whether tomographic score is successful or not in different body mass index groups?

SECONDARY OUTCOMES:
Hospitalization days of the patients according to body mass index groups? | Within a month
  If a patient hospitalized in the clinical ward, how many days the patients hospitalized in the clinic. Grouped as less than 10 days or more than 11 days.
Need for intensive care unit hospitalization | Within a month
  If the patient has a severe course of acute pancreatitis (those with organ insufficiency lasting more than 48h. (such as lung, gastrointestinal system, kidney, etc), the patient is hospitalised into the intensive care unit. Marked as yes or no.
Did the patient lose his life due to AP? | Within a month
  The patient may be alive or may be died because of the acute pancreatitis.
Whether interventional procedures such as endosonography or endoscopic retrograde cholangiopancreatography are required due to the patient's disease | Within a month
  If patients have choledochal stone or cholangitis or micro stones, some interventions may needed such as endosonography or endoscopic retrograde cholangiopancreatography. Need of this procedures marked as yes or no.
How many times has the patient had an acute pancreatitis attack? | Through study completion, an average of 1 year
  Some patients may have several acute pancreatitis attacks; 2,3,4 etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ali̇ Tüzün Ince, Principal Investigator — Bezmialem Vakif Universitesi
Locations (1):
- Bezmialem Vakif University, Gastroenterology Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Result] Khatua B, El-Kurdi B, Singh VP. Obesity and pancreatitis. Curr Opin Gastroenterol. 2017 Sep;33(5):374-382. doi: 10.1097/MOG.0000000000000386. PMID 28719397
- [Result] Shin KY, Lee WS, Chung DW, Heo J, Jung MK, Tak WY, Kweon YO, Cho CM. Influence of obesity on the severity and clinical outcome of acute pancreatitis. Gut Liver. 2011 Sep;5(3):335-9. doi: 10.5009/gnl.2011.5.3.335. Epub 2011 Aug 18. PMID 21927663
- See also: Prevalence of overweight among adults, BMI >= 25 (age-standardized estimate) (%) — https://www.who.int/data/gho/data/indicators/indicator-details/GHO/prevalence-of-overweight-among-adults-bmi-=-25-(age-standardized-estimate)-(-)
- See also: Prevalence of obesity among adults, BMI >= 30 (crude estimate) (%) — https://www.who.int/data/gho/data/indicators/indicator-details/GHO/prevalence-of-obesity-among-adults-bmi-=-30-(crude-estimate)-(-)